CLINICAL TRIAL: NCT00772746
Title: Effectiveness of Specific Model of Cognitive-Behavioral Therapy in Panic Disorder Patients With Agoraphobia
Brief Title: Cognitive Behavioral Therapy in Panic Disorder
Acronym: CBT
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Antonio Egidio Nardi, Universidade Federal do Rio de Janeiro
Other Study IDs: ALSK 021; ALK-123456-1
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Panic Disorder
Keywords: panic; respiration; anxiety; exercise; cognition
MeSH Terms: conditions — Panic Disorder; Respiratory Aspiration; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — None retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- exercise: Respiratory and cognitive exercises in panic disorder patients.

SUMMARY:
The investigators hypothesized that the group of patients receiving the medication interventions and CBT would show significant changes in their behavior, such as remission or reduction in anxiety, panic attacks, anticipatory anxiety, fear of body sensations, loss of control, and agoraphobia avoidance. And also, in the general evaluation of well-being, in the beginning and end of the treatment, in comparison to the control group (medication without CBT), during the same period.

DETAILED DESCRIPTION:
This trial consisted in tracing the profile and evaluating their response to cognitive-behavioral techniques in a sample of 50 panic disorder patients with agoraphobia treated at the Psychiatric Institute of the Federal University of Rio de Janeiro/Brazil. Objective: To test a specific model of cognitive-behavioral therapy through instruments applied in the beginning and end of the procedures. Two groups of 25 patients were formed, the first one with medication and therapy and the second one with medication and without therapy, as the control group. Methods: The cognitive-behavioral therapy sessions were held weekly and individually, with one-hour sessions. The work focused on physiological, cognitive and behavioral aspects with techniques of cognitive reorganization, exercises of induction of symptoms, "in vivo" exposure, breathing and relaxation exercises. The prescribed medication consists of tricyclic antidepressants (TCA) or selective serotonin reuptake inhibitors (SSRI). Results: There was a significant difference between the initial and final evaluation of the group with the specific therapy, such as, reduction in panic attacks, anticipatory anxiety, agoraphobia avoidance, and fear of body sensations. In the global assessment functioning scale, global well-being increased from 60.8% to 72.5% among patients in the first group with therapy, differently from the group without therapy. We observed that 77.6% of the sample in both groups presented the respiratory subtype and 22.4% the non-respiratory subtype. Conclusion: The association of specific cognitive-behavioral therapy focusing on somatic complaints associated with pharmacologic treatment in the first group was effective in this sample, in comparison to pharmacological treatment alone in panic disorder patients with agoraphobia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Both genders with a diagnosis of panic disorder and agoraphobia without severe comorbidities.

Exclusion Criteria:

* Patients showing alcohol or drug dependence
* Mental retardation
* Any other severe mental disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: panic disoder patients over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Beck anxiety inventory Sheehan disability scale fear and phobia questionnaire agoraphobia cognitions questionnaire panic and agoraphobia scale mobility inventory | for observational studies

SECONDARY OUTCOMES:
Beck anxiety inventory Sheehan disability scale fear and phobia questionnaire agoraphobia cognitions questionnaire panic and agoraphobia scale mobility inventory | for observational studies

CONTACTS AND LOCATIONS:
Overall Officials: Antonio E Nardi, MD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- See also: Related Info — http://www.ipub.ufrj.br